CLINICAL TRIAL: NCT02570971
Title: Mannitol Versus Supportive Care in Ciguatera Fish Poisoning: A Randomized Control Trial
Brief Title: Mannitol Versus Supportive Care in Ciguatera Fish Poisoning
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of South Florida (Other)
Collaborators: Florida Poison Control Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CITX-2015
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Ciguatoxin
Keywords: mannitol; treatment
MeSH Terms: interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Control (No Intervention): Patients will receive supportive care measures.
- Investigational (Experimental): Patients will receive 500mL of 20% mannitol
  Interventions: Drug: Mannitol

INTERVENTIONS:
Drug: Mannitol
  Arms: Investigational

SUMMARY:
Ciguatera poisoning, caused by the ingestion of ciguatoxin-containing fish, is a global public health concern. In the US, the vast majority of ciguatera poisonings occur in Florida, followed by Hawaii and California. Equipoise exists in the medical literature regarding the effectiveness of mannitol therapy in treatment of ciguatera poisoning. While there are many case reports attesting to its utility, the only randomized control trial (RCT) comparing mannitol therapy with supportive care failed to show any significant benefit from mannitol treatment for a variety of clinical outcomes. Investigators therefore propose a second, larger RCT to test this question.

ELIGIBILITY:
Inclusion Criteria:

* History consistent with ciguatera poisoning

Exclusion Criteria:

* Minors
* pregnant patients
* those unable to give consent
* severe congestive heart failure or renal failure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Symptom score | 24 hours
  Covers a variety of neurological and gastrointestinal symptoms on a 0-4 score